CLINICAL TRIAL: NCT01699243
Title: A Continuous, Noninvasive Method for Estimating and Predicting Maternal and Fetal Hemodynamic Changes During Regional Anesthesia
Brief Title: Continuous Noninvasive Method for Estimating and Predicting Maternal and Fetal Hemodynamic Changes During Regional Anesthesia
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 12-0990
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Pregnancy; Anesthesia
Keywords: pregnancy; labor; epidural; fetal intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Epidural: subjects under epidural anesthesia

SUMMARY:
Machine learning techniques and algorithms originally developed for use in the field of robotics can be applied to continuous, noninvasive physiological waveform data to discover hidden, hemodynamic relationships. Newly developed algorithms can, in real-time: 1) predict cardiovascular collapse well ahead of any clinically significant changes in standard vital signs, 2) monitor and estimate fluid resuscitation needs, 3) estimate acute blood loss volume, and 4) estimate intracranial pressure. The investigators hypothesize that these same methods can be used to predict functional hypovolemia during regional anesthesia for labor or fetal intervention.

DETAILED DESCRIPTION:
Specific aims:

1. Collect noninvasive physiological waveform data from patients undergoing regional anesthesia for labor or fetal intervention at the University of Colorado Hospital and Children's Hospital Colorado.
2. Combine the physiological data from patient monitors with clinical and demographic data, including maternal problem list, medications, volume infused, use of vasopressors, arterial and venous pressures, fetal heart rate, fetal umbilical artery Doppler velocimetry, maternal uterine artery Doppler waveform, fetal and neonatal outcomes etc. for use in developing mathematical model for early detection of maternal functional hypovolemia.
3. Develop robust, real-time, computational models for:

   * estimating maternal volume status prior to administration of epidural anesthesia
   * estimating effective intravascular volume loss during maternal regional anesthesia
   * predicting an optimal, individual specific requirement for IV resuscitation and/or need for vasopressor agents while providing adequate analgesia using regional techniques and optimizing the fetal outcomes
   * identifying mothers susceptible to epidural induced hypotension

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 14 - 44 years
* 2. Pregnant
* 3. Undergoing regional anesthesia for labor or fetal intervention at the University of Colorado Hospital and Children's Hospital Colorado

Exclusion Criteria:

* 1. Severe pre-eclampsia/eclampsia
* 2. Pre-procedural maternal hypertension requiring treatment
* 3. Significant fetal heart rate abnormalities prior to regional anesthesia
* 4. Incarcerated
* 5. Decisionally challenged
* 6. Limited access to or compromised monitoring sites for non-invasive finger and ear or forehead sensors

Ages: 14 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pregnant females undergoing regional anesthesia for labor or fetal intervention at the University of Colorado Hospital and Children's Hospital Colorado.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
effective intravascular volume loss during maternal regional anesthesia | during epidural, 1-4 hours
  Develop algorithm for estimating effective intravascular volume loss during maternal regional anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Steve Moulton, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado